CLINICAL TRIAL: NCT04252781
Title: Incident Chronic Obstructive pulmoNary dIsease Cohort Study (ICONIC)
Acronym: ICONIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K180305J
Record Dates: First submitted 2020-01-06; First posted 2020-02-05 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Smokers; Chronic Obstructive Pulmonary Disease
Keywords: Incident Chronic Obstructive Pulmonary Disease; comorbidities; trajectories
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exhaustive exploration (Other): Exhaustive exploration of newly diagnosed COPD patients (pulmonary pathology and associated comorbidities)
  Interventions: Other: Exhaustive exploration

INTERVENTIONS:
Other: Exhaustive exploration — * clinical investigations
  * imagery
  * blood assessment
  * functional respiratory investigations
  * muscle function / skeletal muscle index

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD), , secondary to smoking, is a major public health issue with very high direct and indirect costs. The impact on the health system of undiagnosed patients, up to 70% of patients, is increasingly documented. However, systematic spirometry screening remains controversial among smokers in the absence of data to link the detection of new patients with improved management and clinical events and health goals. More generally, there is little data on the evolution of patients in real life once they have entered the care system.

The premise is that with systematic screening in general medicine, it is possible to identify the evolution of newly diagnosed COPD patients, to distinguish the different possible evolutions according to the initial phenotype and the management.

DETAILED DESCRIPTION:
A description of the population from which the groups or cohorts will be selected Smokers who have a screening spirometry for COPD, either in general medicine, at a pulmonologist or in the CHIC or Henri Mondor hospital respiratory function tests department.

After screening, an equal number of men and women COPD will be included (150 men and 150 women). 1500 smokers will be included to reach 300 smokers with COPD.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of smokers with spirometry (pre-inclusion)

* Age> 35 years
* Smoking > 20 PA
* Active smoking (cessation < 1 month)
* Signature of consent to participate in Phase I of the study

Inclusion criteria for patients with incidental COPD

* FEV1 / FVC <70% of the theoretical value and / or <LLN (Lower limit of normal)
* Signature of consent to participate in Phase II of the study

Exclusion Criteria:

* Known COPD
* Cancer being treated
* No affiliation to the social security or other social protection scheme
* Pregnant or lactating woman
* Patient deprived of liberty or under legal protection (under tutorship or curatorship

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — After screening, an equal number of men and women COPD will be included (91 men and 92 women).
Enrollment: 300 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
1-year adverse evolution | at 12 Months
  1-year adverse evolution defined by a composite criterion associating:
  - Occurrence of an additional exacerbation defined by any event requiring the use of the care system (visit to the doctor, emergencies, or hospitalization, for respiratory aggravation) with prescription of antibiotics or systemic steroids
  AND/OR
  - Increased dyspnea by 1 point on the MMRC dyspnea score
  AND/OR
  - CAT> 10 or 2 points increase on CAT symptom scores

SECONDARY OUTCOMES:
Adverse evolution | at 3 Months and 6 Months
  - Occurrence of an additional exacerbation defined by any event requiring the use of the care system (visit to the doctor, emergencies, or hospitalization, for respiratory aggravation) with prescription of antibiotics or systemic steroids
  AND/OR
  - Increased dyspnea by 1 point on the MMRC dyspnea score
  AND/OR
  - CAT> 10 or 2 points increase on CAT symptom scores
Exacerbation | at 3 Months, 6 Months and 12 Months
  Occurrence of an additional exacerbation defined by any event requiring the use of the care system (visit to the doctor, emergencies, or hospitalization, for respiratory aggravation) with prescription of antibiotics or systemic steroids
Number of steps | at 3 Months, 6 Months and 12 Months
  Number of steps in the month preceding the visit evaluated by a pedometer
Forced Expiratory Volume in one second (FEV1) | at 3 Months, 6 Months and 12 Months
  Forced Expiratory Volume in one second (FEV1)
Hospital Anxiety and Depression scale | at 3 Months, 6 Months and 12 Months
  Anxious symptoms or depressions
FEV 1 / Respiratory function parameters | at 12 Months
  Respiratory function parameters with FEV 1
DLCO / Respiratory function parameters | at 12 Months
  Respiratory function parameters with DLCO
Residual volume / Respiratory function parameters | at 12 Months
  Respiratory function parameters with residual volume
Total lung capacity / Respiratory function parameters | at 12 Months
  Respiratory function parameters with total lung capacity
Arterial stiffness | at 12 Months
  Arterial stiffness measured by the pulse wave velocity (Complior)
LVEF / Echocardiography | at 12 Months
  LVEF measured by echocardiography
Diastolic dysfunction / Echocardiography | at 12 Months
  diastolic dysfunction measured by echocardiography
PAPS / Echocardiography | at 12 Months
  PAPS measured by echocardiography
Skeletal muscle index | at 12 Months
  Skeletal muscle index evaluated by IDEXA
Muscle function | at 12 Months
  Muscle strength by grip and pinch
Hospital Anxiety and Depression scale | at 12 Months
  Measurement of anxiety symptoms or depression via the Hospital Anxiety and Depression scale.
Numbers of deaths | at 12 Months
  Numbers of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BOYER, MD, Principal Investigator — Assistance Publique Hôpitaux de Paris (AP-HP)
Locations (1):
- Hopital Henri MONDOR, Créteil, Île-de-France Region, France